CLINICAL TRIAL: NCT06966895
Title: The Effectiveness of Parent-child Collaborative Game on Children Attentiveness in Informal Learning Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhu Dian, Dr, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NEADS005
Record Dates: First submitted 2024-09-01; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-09

CONDITIONS: Education; Educational Technology; Children; Knowledge
Keywords: informal learning environment; attentiveness; parent-child collaboration; game

STUDY DESIGN:
Intervention Model Description: In terms of user motivation, the gamified design model for museums aims to engage and satisfy both parents and children by tapping into their intrinsic and extrinsic motivations. The goal is to enhance their involvement and enjoyment. The model emphasizes social interaction and curiosity, offering opportunities for enjoyment and a sense of accomplishment through interactions with parents and peers. By incorporating game-like challenges, the model caters to children&#39;s natural inclination for exploration, igniting their curiosity and thus increasing their interest and engagement with the museum.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Museum Talking (Experimental): This application is utilized throughout the entire behavioral process of a museum visit; it serves as an auxiliary tool to facilitate the parent-child groups' experience in the museum in a more targeted manner. The players will experience the historical narrative, Breakout Q&A,and the production game in collaboration with parents. Players can earn between 0 and 3 stars in the game, contingent on the frequency of accurate responses.While the breakout mechanism is mainly triggered by children's external motivation, the design parts of the internal motivation are mainly triggered by parental involvement, including the APP hints, and the model kitchen game. During the first two levels of answering questions, parents get some hints through the APP. In the third level of the simulated kitchen, parents get detailed cooking recipes through the APP so that children can finish it with the help of their parents. The simulated kitchen is a real space containing plastic cookware and ing
  Interventions: Device: a parent-child collaboration game app
- Traditional text-based panels group (Sham Comparator): A traditional museum visitor's manual, containing knowledge of similar content to that in the game.
  Interventions: Other: traditional text-based panels group

INTERVENTIONS:
Device: a parent-child collaboration game app — This application is utilized throughout the entire behavioral process of a museum visit; it serves as an auxiliary tool to facilitate the parent-child groups' experience in the museum in a more targeted manner.
  Arms: Museum Talking
Other: traditional text-based panels group — A traditional museum visitor's manual, containing knowledge of similar content to that in the game.
  Arms: Traditional text-based panels group

SUMMARY:
To assess the impact of applying a parent-child collaboration game app on children during museum visiting process compared to traditional text-based panels.

DETAILED DESCRIPTION:
The objective of our research was to confirm the efficacy of an interactive app that facilitates parent-child collaboration during museum visits and to provide children with knowledge regarding the museum learning process. An application is utilized throughout the entire behavioral process of a museum visit; it serves as an auxiliary tool to facilitate the parent-child experience in the museum in a more targeted manner.

ELIGIBILITY:
Inclusion Criteria:

1. age 8-10 years,
2. good communication and comprehension skills without significant cognitive deficits
3. parents' ability to operate electronic devices proficiently.

Exclusion Criteria:

1. children can't read the text accurately
2. children with severe disabilities who are unable to move easily
3. guardians who are responsible for more than one child

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
FSS (Flow State Scale) score | immediately after the procedure
  The Flow State Scale (FSS) is a psychological assessment tool used to measure the experience of flow, a state of deep immersion and focus in an activity, where time seems to disappear, and a person feels fully engaged and in control. Flow is often associated with peak performance in various domains, including sports, work, and creative activities.
  The FSS typically consists of a series of statements related to the nine dimensions of flow (Challenge-Skill Balance, Action-Awareness Merging, Clear Goals, Unambiguous Feedback, Concentration on the Task, Sense of Control, Loss of Self-Consciousness, Transformation of Time and Autotelic Experience).
  Respondents typically rate each statement on a Likert scale (e.g., from 1 to 5 or 1 to 7), indicating how much they agree or disagree with each statement as it applies to their experience. Higher scores on the FSS indicate a stronger experience of flow.

SECONDARY OUTCOMES:
Post-game knowledge assessment | immediately after the procedure
  The Knowledge Test was designed to analyze educational efficiency by measuring the amount of knowledge remembered by participants. The test consisted of seven quiz questions about points of knowledge in the museum. In order to prevent children from visiting purposefully, the researcher designed two similar sets of test questions.

CONTACTS AND LOCATIONS:
Overall Officials: Dian Zhu, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Information concerning children